CLINICAL TRIAL: NCT06384170
Title: Closed Loop Spinal Cord Stimulation (SCS) for Neuromodulation of UMN-Lesion Spasticity
Brief Title: Closed Loop Spinal Cord Stimulation for Neuromodulation of Upper Motor Neuron Lesion Spasticity
Acronym: CLONUS
Status: Withdrawn | Type: Observational
Why Stopped: The study will not move forward; lack of staff
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00442113
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain; Spasticity as Sequela of Stroke; Upper Motor Neuron Lesion
Keywords: Spinal Cord Stimulation; Neuromodulation; Closed-loop SCS; Post-Stroke Pain; Spasticity; Chronic Pain; Functional Recovery
MeSH Terms: conditions — Chronic Pain; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Interventional: Patients identified with post-stroke pain due to spasticity. Patients will be evaluated for spinal cord stimulation trial. The trial will be for 7 days.
  Interventions: Device: Spinal Cord Stimulation- Closed loop

INTERVENTIONS:
Device: Spinal Cord Stimulation- Closed loop — This is a percutaneously placed epidural electrode that is connected to a battery-powered impulse generator for power. The electrical delivery is monitored in real-time with the measurement of evoked compound action potentials and adjusted to provide titration of therapeutic stimulation delivery.

SUMMARY:
Spasticity is characterized by increased muscle tension and is a classic consequence of upper motor neuron (UMN) damage in the central nervous system, such as from stroke or trauma. Clinically, it presents as muscle resistance to passive stretching, along with clasp-knife rigidity, clonus, increased tendon reflexes, and muscle spasms. An imbalance of the descending inhibitory and muscle stretch reflexes is thought to be the cause of spasticity. Post-stroke spasticity is a common condition that occurs in 37.5-45% of cases in the acute stage and 19-57.4% in the subacute stage after a stroke. At 6 months post-stroke, spasticity develops in 42.6-49.5% of cases, and at one year, it affects 35-57.4% of individuals. In patients with cerebral palsy (CP), incidence is almost 80% while in those living with spinal cord injury the number approaches up to 93%. Traumatic brain injury (TBI) patients have a higher prevalence on initial admission to neurorehabilitation but one in three patients will have chronic spasticity. However, the Defense and Veterans Brain Injury Center report a rate of TBIs amongst deployed veterans to be around 11-23% mostly from blast and explosive trauma.

There have been studies as early as the 1980s exploring the efficacy of SCS for spasticity control, however, the credibility of many of these studies is constrained due to an incomplete comprehension of spasticity's underlying mechanisms, outdated research methods, and early limitations in implantable device technology. Intrathecal pumps for baclofen have remained as the mainstay for refractory spasticity, however, it comes with associated risks such as chemical dependence leading to acute baclofen withdrawal and requiring frequent refill requirement. Most importantly, it does not yield functional improvement of muscle activity, just suppression of spasticity. Botox is also routinely used but due to heterogeneity in muscle involvement as well as variability in provider skill, results may be inconsistent and short-lasting, requiring frequent clinic visits for repeat injections to the affected muscle groups. SCS may be able to address that gap in spasticity management.

ELIGIBILITY:
Inclusion Criteria:

1. First-ever stroke
2. Aged 18 and older
3. Neuropathic pain >3 months (chronic)
4. Brain injury associated with spasticity in one or multiple limbs >3 months post-stroke
5. No previous history of neuropathic pain or spasticity in affected limbs
6. Cognitively capable to operate the SCS system

Exclusion Criteria:

1. Inadequate Pain Severity: Patients with mild or non-debilitating pain may be excluded if the treatment is intended for individuals with moderate to severe pain.
2. Previous SCS Implantation: Patients who have previously undergone SCS implantation may be excluded to focus on those who are new to the therapy.
3. Inadequate Pain Duration: Some trials may exclude patients whose pain has not persisted for a minimum period to ensure that the pain condition is chronic.
4. Medical Comorbidities: Patients with certain medical conditions or comorbidities that may increase the risks associated with SCS, such as uncontrolled cardiovascular disease, uncontrolled diabetes, or active infections, may be excluded.
5. Psychological Factors: Patients with severe psychiatric disorders or psychological conditions that may interfere with the assessment of pain or the ability to provide informed consent may be excluded.
6. Allergies or Sensitivities: Patients with allergies to materials used in SCS devices or contraindications to the anesthesia used during implantation may be excluded.
7. Substance Abuse: Patients with active substance abuse or addiction issues may be excluded due to concerns about treatment compliance and efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A subject who meets all of the inclusion criteria, and none of the exclusion criteria, is eligible to participate in the study. A subject is considered enrolled when the subject signs the subject informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Pain as assessed by Visual Analog Score | baseline (pre-procedure), day 1 (post-procedure) day 7 (trial lead removal), day 14 (7 days post removal)
  Visual Analog Scores, pain score with possible range from zero (no pain) to ten (worst imaginable pain)

SECONDARY OUTCOMES:
Spasticity Reduction as assessed by the Modified Ashworth's Score | baseline (pre-procedure), day 1 (post-procedure) day 7 (trial lead removal), day 14 (7 days post removal)
  Modified Ashworth's Scores range from 0-4. Minimum score is '0' meaning no increase in tone. Maximum score is '4' meaning limb is ridged in flexion and extension. The lower the score the better the outcome
Short Form 36 Health Survey (SF-36) score | baseline (pre-procedure), day 1 (post-procedure) day 7 (trial lead removal), day 14 (7 days post removal)
  The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. The total score on the SF-36 ranges from 0 - 100 Lower scores = more disability, higher scores = less disability
Medication Use | baseline (pre-procedure), day 1 (post-procedure) day 7 (trial lead removal), day 14 (7 days post removal)
  Dose and frequency of medication use for current symptoms
Health Status as assessed by the EuroQol 5 Dimension 5 Level (EQ-5D-5L) | baseline (pre-procedure), day 1 (post-procedure) day 7 (trial lead removal), day 14 (7 days post removal)
  Effects on health-related quality of life that comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The survey is scored in two separate sections. The first section is measured by a minimum score of 5 and a maximum score of 25. Higher score greater level of problems. The second section measures self report health status on a 0 to 100. Higher score best health.

OTHER OUTCOMES:
Spinal cord neurophysiological wave morphology | day 1 (post-procedure), continuous data capture until day 7 (or until trial lead removal), day 14 (7 days post removal)
  Assessed using data downloaded from the implanted closed-loop SCS system. Will measure and report on the various morphologies of the Evoked Compound Action Potentials (ECAPs).
Spinal cord neurophysiological Current (mA/mV) | day 1 (post-procedure), continuous data capture until day 7 (or until trial lead removal), day 14 (7 days post removal)
  Assessed using data downloaded from the implanted closed-loop SCS system. Will measure and report on the current (mA/mV) of the Evoked Compound Action Potentials (ECAPs).
Spinal Cord Neurophysiological Characteristic- Conduction Velocity (m/s) | day 1 (post-procedure), continuous data capture until day 7 (or until trial lead removal), day 14 (7 days post removal)
  Assessed using data downloaded from the implanted closed-loop SCS system. Will measure and report on the conduction velocity (m/s) of the Evoked Compound Action Potentials (ECAPs).

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Chhatre, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayorova L, Radutnaya M, Varyukhina M, Vorobyev A, Zhdanov V, Petrova M, Grechko A. Immediate Effects of Anti-Spastic Epidural Cervical Spinal Cord Stimulation on Functional Connectivity of the Central Motor System in Patients with Stroke- and Traumatic Brain Injury-Induced Spasticity: A Pilot Resting-State Functional Magnetic Resonance Imaging Study. Biomedicines. 2023 Aug 14;11(8):2266. doi: 10.3390/biomedicines11082266. PMID 37626762
- [Background] Powell MP, Verma N, Sorensen E, Carranza E, Boos A, Fields DP, Roy S, Ensel S, Barra B, Balzer J, Goldsmith J, Friedlander RM, Wittenberg GF, Fisher LE, Krakauer JW, Gerszten PC, Pirondini E, Weber DJ, Capogrosso M. Epidural stimulation of the cervical spinal cord for post-stroke upper-limb paresis. Nat Med. 2023 Mar;29(3):689-699. doi: 10.1038/s41591-022-02202-6. Epub 2023 Feb 20. PMID 36807682
- [Derived] Abstracts of Scientific Papers and Posters Presented at Physiatry '25: February 25 - March 1, 2025. Am J Phys Med Rehabil. 2025 Jun 1;104(6S Suppl 1):S1-S240. doi: 10.1097/PHM.0000000000002746. No abstract available. PMID 40421840